# Statistical Analysis Plan

Protocol No. MT-1186-J06
Clinical Pharmacology Study of Oral Edaravone in Healthy Adult Subjects
(Food Effect Study)

| Prepared By: | Mitsubishi Tanabe Pharma Corporation |
|--------------|--------------------------------------|
| Version: | Version 1.0 |
| Date: | 28Nov2019 |

NCT number: NCT05342597

# APPROVAL FORM Statistical Analysis Plan

| Protocol No. | MT-1186-J06 |
|---|---|
| Protocol Title | Clinical Pharmacology Study of Oral Edaravone in Healthy Adult |
| | Subjects (Food Effect Study) |
| Version / Date | Version 1.0/ |

# Authors:

| Statistics Author | |
|-------------------|------------------|
| Print Name: | |
| Position: | COT STAT |
| Clinical Pharmac | okinetics Author |
| Print Name: | |
| Position: | COT CP |

| Approved by: | |
|---------------------|------------------|
| Statistic Approver | |
| Print Name: | |
| Position: | Responsible STAT |
| Signature: | |
| Approval date: | |
| Clinical Pharmacoki | netic Approver |
| Print Name: | |
| Position: | Responsible CP |
| Signature: | |
| Approval date: | |

# TABLE OF CONTENTS

| 1. | INTRODUCTION | 7 |
|---|---|---|
| 2. | STUDY OBJECTIVE AND ENDPOINTS | 7 |
| | 2.1. Study Objectives | 7<br>7 |
| 3. | STUDY DESIGN | 7 |
| | 3.1. Phase and Type of the Study | 8<br>8<br>8<br>9 |
| 4. | PLANNED ANALYSIS | 3 |
| | 4.1. Final Analysis | |
| 5. | ANALYSIS POPULATIONS | 4 |
| 6. | STATISTICAL CONSIDERATIONS1 | 4 |
| | 6.1. Descriptive Statistics16.2. Statistical Tests16.3. Data Review Meeting1 | 4 |
| 7. | DATA CONVENTIONS | 5 |
| | 7.1. Analysis Variable Definitions 1 7.1.1. Study Subjects 1 7.1.1.1. Demographic and Other Baseline Characteristics 1 7.1.1.2. Medical History 1 7.1.1.3. Prior or Concomitant Medication 1 7.1.2. Safety Assessments 1 7.1.2.1. Adverse Events 1 7.1.2.2. Laboratory Tests 1 7.1.2.3. 12-Lead ECG 1 7.1.3. Pharmacokinetics Evaluation 1 7.1.3.2. Pharmacokinetic Parameters 1 7.2. Analysis Visit Definitions 1 7.3. Data Handling Convention for Missing Data 2 | 5<br>5<br>5<br>5<br>6<br>6<br>8<br>8<br>8<br>8<br>8<br>9<br>20 |
| 8. | STATISTICAL METHODOLOGY2 | |
| | 8.1. Study Subjects | 20<br>20<br>20 |

| | 8.1.5. Medical History and Allergic History21 |
|---|---|
| | 8.1.6. Prior or Concomitant Medications |
| | 8.2. Efficacy Assessments |
| | 8.3. Safety Assessments |
| | 8.3.1. Adverse Events |
| | 8.3.2. Laboratory Tests |
| | 8.3.3. Vital Signs |
| | 8.3.4. 12-Lead ECGs |
| | 8.3.5. Physical Examinations |
| | 8.4. Pharmacokinetics Evaluation |
| | 8.4.1. Concentrations and Pharmacokinetic Parameters for unchanged edaravone, sulfate conjugate, and glucuronide conjugate 24 |
| | 8.4.2. Analysis of Food Effect |
| 9. | DATA PRESENTATION CONVENTIONS25 |
| | 9.1. Number of Digits to Report |
| | 9.2. Treatments to Report |
| | 9.3. Analysis Visits to Report |
| 10. | CHANGE FROM THE PROTOCOL27 |
| 11. | SOFTWARE |
| 12. | REFERENCES27 |

# **ABBREVIATIONS**

| Abbreviations | Definitions |
|---------------|----------------------------------------------|
| AE | adverse event |
| ALT | alanine transaminase |
| ALP | alkaline phosphatase |
| AST | aspartate transaminase |
| ATC | anatomical therapeutic chemical |
| BLQ | below limit of quantification |
| BMI | body mass index |
| CI | confidence interval |
| CV | coefficient of variation |
| DP | decimal places |
| DRM | data review meeting |
| ECG | electrocardiogram |
| MedDRA | medical dictionary for regulatory activities |
| PK | pharmacokinetics |
| PT | preferred term |
| SAP | statistical analysis plan |
| SAE | serious adverse event |
| SAF | safety population |
| SD | standard deviation |
| SOC | system organ class |
| WHO | World Health Organization |

# LIST OF PK PARAMETERS

| Parameters | Definitions |
|---|---|
| AUC <sub>0-24</sub> | Area under the plasma concentration-time curve from zero up to 24 hour |
| AUC <sub>0-t</sub> | Area under the plasma concentration-time curve from zero up to the last quantifiable concentration time point |
| AUC₀-∞ | Area under the plasma concentration-time curve from zero up to infinity with extrapolation of the terminal phase |
| AUC% <sub>ex</sub> | Area under the (plasma) concentration-time curve extrapolated from the last |
| | quantifiable concentration time point to infinity in % of the total AUC₀-∞ |
| Ae <sub>0-24</sub> | Cumulative urinary excretion amount of drug from zero to 24 hour |
| Ae <sub>0-48</sub> | Cumulative urinary excretion amount of drug from zero to 48 hour |
| C <sub>max</sub> | Maximum plasma concentration after administration |
| C <sub>last</sub> | Last quantifiable concentration |
| CL/F | Apparent total clearance |
| CLr | Renal clearance |
| Kel | Elimination rate constant from the central compartment |
| LLOQ | Lower limit of quantification |
| LOQ | Limit of quantification |
| MRT | Mean residence time |
| NC | Not calculated |
| t <sub>1/2</sub> | Terminal elimination half-life in plasma concentration-time course |
| V <sub>ss</sub> /F | Apparent volume of distribution at steady state |
| V <sub>z</sub> /F | Apparent volume of distribution during terminal phase |
| Ae% | Urinary excretion ratio of drug |

#### 1. INTRODUCTION

This statistical analysis plan (SAP) is based on the final protocol (v1.0) dated 13-May-2019. The plan covers statistical analysis, tabulations and listings of the study data to investigate the pharmacokinetics (PK) and safety.

The SAP is prepared by Mitsubishi Tanabe Pharma Corporation (MTPC). The statistical analysis and production of the outputs described in the SAP and QC will be conducted by . The final analysis and outputs will be checked by

and approved by MTPC Data Science Department.

Any statistical analysis details described in this document supersede any description of statistical analysis in the protocol.

#### 2. STUDY OBJECTIVE AND ENDPOINTS

2.1. Study Objectives

Primary objective: To evaluate the effect of food on the PK of oral edaravone in healthy

adult subjects.

Secondary objective: To evaluate the PK, safety, and tolerability of oral edaravone.

#### 2.2. Study Endopoints

# 2.2.1. Safety Assessments

- (1) Adverse events and adverse drug reactions
- (2) 12-lead ECG
- (3) Laboratory tests
- (4) Vital signs

# 2.2.2. Pharmacokinetics Assessments

(1) Drug concentration (in plasma and urine)
Unchanged edaravone, sulfate conjugate, and glucuronide conjugate

(2) Pharmacokinetic parameters

Unchanged edaravone:  $AUC_{0-24}$ ,  $AUC_{0-t}$ ,  $AUC_{0-\infty}$ ,  $C_{max}$ ,  $t_{max}$ ,  $t_{1/2}$ , Kel, MRT, CL/F,  $V_z/F$ ,  $V_{ss}/F$ , Ae, Ae%, CLr

Sulfate conjugate and glucuronide conjugate:  $AUC_{0-t}$ ,  $AUC_{0-24}$ ,  $AUC_{0-\infty}$ ,  $C_{max}$ ,  $t_{max}$ ,  $t_{1/2}$ , Kel, Ae, Ae% (t: Final concentration measurable time point)

Other PK parameters (for all PK profiles for which the Kel has been calculated): AUC%<sub>ex</sub>, Adjusted R<sup>2</sup>, Number of Kel points, Lower limited of Kel, Upper limiter of Kel

#### 3. STUDY DESIGN

# 3.1. Phase and Type of the Study

Phase of the study: Phase I

Type of the study: Clinical pharmacology study

# 3.2. Study Design

# 3.2.1. Type and Details of Cohorts

Single-dose, randomization, open-label, crossover study

| | | , | · | | |
|---|---|---|---|---|---|
| Group | Period I<br>(at Day 1) | Period II<br>(at Day 3) | Period III<br>(at Day 5) | Period IV<br>(at Day 7) | Period V<br>(at Day X+1) |
| 1 | Α | В | С | D | The diet condition will |
| 2 | В | C | D | A | be determined based on<br>the PK data collected |
| 3 | С | D | A | В | from period I to period IV. *) |
| 4 | D | Α | В | С | (E, F, or G etc.) |

- A: Dosing under fasted condition
- B: Dosing 8 hours after high-fat meal
- C: Dosing 4 hours after low-fat meal
- D: Dosing 2 hours after light meal
- \*) The diet menu (any one of high-fat meal, low-fat meal and light meal) and dosing time after a meal (within a range of 30 minutes to 10 hours after a meal) in period V will be determined based on the PK data collected from period I to period IV. The possible case of the diet condition includes the following.
- E: Dosing 2 hours after low-fat meal
- F: Dosing 4 hours after light meal
- G: Dosing 8 hours after low-fat meal



#### 3.2.2. Study Period and Evaluation Period

Study period: The study period is defined as the period from the time of obtaining the informed consent to the time of completion of the end-of-study assessment or discontinuation assessment (for subjects who have entered into the follow-up period, to the time of completion or termination of the follow-up).

Screening: Subjects providing informed consent will be screened for eligibility to select subjects meeting all of the inclusion criteria and none of the exclusion criteria (16 subjects with a few reserve subjects).

Evaluation period: The evaluation period is defined as the period from completion of dosing of the investigational product on Day 1 to completion of the end-of-study assessment or discontinuation assessment. The duration of hospitalization will be 10 days and 9 nights

(Day -1 to Day 9) for Period I to Period IV, and 4 days and 3 nights (Day X to Day X+3) for Period V.

End-of-study assessment: The prespecified observations and tests will be performed as the end-of-study assessment, 7 days (±2 days) after the last dose of the investigational product.

# 3.3. Schedule of Study Procedures

| Group 1: Period I to IV | Group | 1: | Pe | riod | Ι | to | $\mathbf{I}$ | 7 |
|-------------------------|-------|----|----|------|---|----|--------------|---|
|-------------------------|-------|----|----|------|---|----|--------------|---|

| | Informed | Screening | | | P | erio | 41( | ΔI | )osi | ag a | ade | T fas | ted | COL | ditie | 20) | | | L | _ | P | s Lio | ш | (B: 1 | Dosi | <b>3</b> 2 | 100 | EC3 2 | đer | أينط | | = | <u>=0</u> | _ | | 4 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day (time window) | consent | Day -30<br>to -2 | -1 | | | | | | | 1 | | | | | | | ⊥ | 2 | | | | | | | _ | 3 | | | | | _ | _ | | ┙ | 4 | |
| Time after doxing | | Visk | Adm ission | Pre-dose | 0 | 5 100 | 15 m | 301 | 458 | 4 | 1 h 30 m | 2.8 | 47 | 4 9 | # | 101 | 17. | 3 2 | 8 h Pre-dose | Pre-dose | 48.5 | 0 | 8 8<br>8 8 | 15 m | 30m | 45m | 41 | 1 b 30 m | 2 h | 4 9 | ч9 | æ | 10 h | 8 21 | 2 2 | 2 |
| Written informed consent | х | | | | | | | | | | | | | | $\Box$ | I | Ι | I | | I | Ι | Ι | Г | | | | | | $\Box$ | | | $\Box$ | $\Box$ | I | ユ | 3 |
| Subject characteristics | T | X | | | | | | | | | | | | | | | | | | $\perp$ | | | L | | L | | | | | _ | | _ | _ | Ц. | _ | |
| Eligibility assessment | | X | X | X | | | | | | | | | | | | | L | | | $\perp$ | I | | L | 匚 | L | L | | | _ | _ | | _ | _ | 4 | _ | |
| Food (High · Low · Light)*) | | | | Г | | | | | | | П | T | | П | [ | | | | Hig | ı | Ι | 1 | | L | | | L | | | | | | | ᆚ | Ш | |
| Dosing of eduratione | 1 | | Г | Г | X | | | | П | | П | | $\neg$ | П | $\perp$ | Т | Ι | | | Τ | Ι | X | | Γ. | | | | | | | | | $\Box$ | $\perp$ | 丄 | |
| Height weight BMIh) | | x | x | Г | | | | Т | | | П | П | T | П | Т | Т | Т | | | Т | Т | Г | Γ | Г | L_ | | | | | | | | | $\perp$ | _L | |
| Physical examination | 1 | X | x | Ī | | | | ┪ | ┑ | x | ┑ | T | | П | 1 | Т | . 12 | K | | 7 | T | $\top$ | Г | | | | X | | | П | | П | | | X | |
| Vital signs | | X | X | X | | Г | | П | П | X | ╗ | T | ┑ | ╗ | Т | Т | 7 | X | Т | 7 | Т | Т. | Г | | | Г | X | | | П | П | | $\Box$ | | X | |
| 12-lead ECG | 1 | x | x | Ī | | | | ┑ | П | X | ヿ | T | $\neg$ | 7 | Т | T | 7 | ĸ | Т | 7 | ī | 1 | Г | | | | X | | | Т | | $\Box$ | $\Box$ | Ŀ | X | |
| Laboraty tests | | x | x | Т | | | | П | | | $\neg$ | | | | $\Box$ | Τ. | Ι | $\perp$ | | Ι | | | | | L | | | | | | | | | ⊥ | | |
| Serological tests | | X | П | | | | | | | | П | Т | _ | П | П | I | | | 1 | Ι | Т | Ц | Г | | L | 匚 | | | | | | | 1 | I | 丄 | |
| Drug/alcohol abuse screening | | x | | Г | | | | П | | | | $\Box$ | | П | $\Box$ | | I | | | I | Т | | | | | | L | | | | | i | | 1 | 丄 | |
| Pregnancy test in female | | X | X | Г | | | | | | | | $\Box$ | | $\Box$ | Ι | Ι | | | I | | Ι | 1 | L | | L | 匚 | L | | | $\Box$ | | $\Box$ | | $\perp$ | ⊥ | |
| Adverse events <sup>a)</sup> | <b>←</b> | | H | F | | | | $\exists$ | | $\exists$ | | $\exists$ | $\exists$ | $\neg$ | $\pm$ | $\pm$ | Ŧ | $\pm$ | <del></del> | Ŧ | $\pm$ | Ε | Ε | Е | E | Е | | | | Ⅎ | <u>∃</u> | $\exists$ | $\exists$ | $\pm$ | $\pm$ | - |
| Concomitant are dications | | < | $\vdash$ | Н | Е | - | | $\exists$ | $\exists$ | $\exists$ | $\equiv$ | $\exists$ | $\exists$ | $\overline{}$ | $\exists$ | $\pm$ | Ŧ | F | $\pm$ | Ξ | Ε | $\pm$ | Е | E | Е | F | Е | Е | | 1 | Ⅎ | $\exists$ | $\exists$ | $\pm$ | $\pm$ | 3 |
| Blood sampling for edaratrone | | | Г | X | | X | X | I | X | X | X | X | xΤ | X | ΣŢ | X : | X : | x x | | $\mathbf{I}$ | 7 | | X | X | X | X | X | X | X | X | X | X | X | XI: | X I | ¢ |
| Urine sampling for educations <sup>d)</sup> | | | Г | 4 | | | П | $\dashv$ | $\exists$ | - | $\neg$ | | $\neg$ | -7 | Ŧ | | = | | = | Ŧ | ┰ | ⇍ | Τ | F | Н | ₽ | F | Ε | - | -7 | -7 | 7 | 7 | Ŧ | Ŧ | ∃ |

| | | | | Peri | od I | II (( | C: D | 05 <u>i</u> | g 4 | bou | T 2 | Rer | low | fut: | mex | ) | | | _ | | | | Per | iod | IV ( | D: 1 | Dosi | | l bo | ars : | Δe | igi | bt 10 | esl) | 1 | | _ | _ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day (time window) | Г | | | | | | | | ; | | | | | | | | | 6 | | | | | | | | | 7 | | | | | | | | ١ | 8 | , | 9 |
| Time after doxing | Before meab | 4 h Pre-dose | Pre-dose | 48 | 0 | 5.0 | 15 m | 30 m | 45 m | 1 | 1 h 30 m | 2.1 | 41 | <b>4</b> 9 | 33 | 10 1 | 12 h | 24 h | 36 h | 2 h Pre-dose | Pre-dose | 46 h | 0 | 5 m | 15 m | 30 m | 45 m | = | 1 h 30 m | 2.6 | 411 | 6 h | 48 | 10 % | 12 k | 24 h | 36 h | Discharge#8 h |
| Written informed consent | t | | t | L | | | | | | | | Ш | | | | | | | | | | | | | | | | | | | | | | | | 口 | ╛ | Ξ |
| Subject characteristics | Г | l''' | T | | | | | | | | | | | | | | | | | | | | | | | | L | L | L | | | | | | ш | ш | | _ |
| Eligibility assessment | Т | | Т | Т | Г | П | | | | | | | | | | | | | | | 1 | | | | | | | | L | | | ш | | | Ш | ш | ┙ | |
| Food (High: Low-Light) <sup>a)</sup> | Т | Low | Т | Т | Г | П | Г | | | Г | | | | | | | | | | Light | | | | | | | | | | L. | | Ш | | | ш | Ш | | |
| Dosing of edaravone | Т | | Т | П | Z | | | | | | | | | | | | | | | | | | Z | | | | | | | L. | | | | | Ш | | | |
| Height, weight, BMI <sup>b)</sup> | Т | | Т | П | Г | | П | | | Г | П | | | | | | | | | | | | | | | Г | Γ | П | | П | | | | | | П | | Г |
| Physical examination | Т | | X | 1 | Т | | Г | | | x | | | П | | Г | | | X | | | X | | | | | | | Z | ľ | | | | | | | Z | | Z, |
| Vital signs | 1 | | Z | Т | Т | | г | | | X | | | П | Г | Г | | | Z | | | Z | | | | | | Т | Z | Г | | | | | Г | | X | | Z |
| 12-lead ECG | т | | 7.7 | Т | Т | - | Г | | | X | | | П | | П | | | X | | | Z | Π. | | | | | Г | Z | | | | | | | | X | | и. |
| Laboraty tests | X | | Т | Т | Г | | Г | | | Г | Т | | П | Г | П | | | | | | Г | | | | | | | Г | Г | | | | | | | | | Z |
| Serological tests | Т | | Τ | Т | Г | | | | | | | | П | | | | | | | | | | | | | | Г | | | | | | | | | | | |
| Drug/alcohol abuse screening | Т | | Т | Т | Г | Г | Π | | | | | | Г | | | | | | | | Π | | | | | | $\Box$ | Г | L | | | | | | | | | |
| Pregnancy test in female | Т | | | Т | П | Τ. | | | | Γ | | | Г | | | | | | | | Π | | | | | | Г | Г | L | | | | | | | | | |
| Adverse events <sup>e)</sup> | k | | Ŧ | ₽ | F | F | | | | F | | F | | | Е | _ | Н | | П | | F | E | Е | - | ł | | ₩ | H | Е | | | oxdot | | - | $\vdash$ | $\Box$ | | Ϊ |
| Concomitant use dications | <b>←</b> | | Ŧ | ₽ | F | F | F | - | | F | | Е | Е | | Е | | | _ | П | | Ε | Ε | | - | ł | | - | Ε | Е | $\equiv$ | $\equiv$ | | | - | | | $\equiv$ | Ϊ |
| Blood sampling for edaravone | 1 | | T | Z | Т | Z | X | X | X | X | X | X | Z | Z | Z | X | Z | Z | X | | | Z | L | X | X | X | X | Ιž | Z | X | Z | Z | X | X | X | X | X | 7 |
| Urine sampling for educations <sup>d)</sup> | k | | 1 | $\rightarrow$ | 1 | = | _ | | | | | | | | Г | _ | | П | П | | Η- | × | | - | Н | Е | - | Н | 1 | Ι | F | | = | Η | | П | | 7 |

- a) High: High-fat meal, Low: Low-fat meal, Light: Light meal
- b) Height will be measured at screening only. Body weight will be measured at screening, admission, and end-ofstudy assessments. BMI will be calculated at screening and admission assessment.
- c) Assess serious adverse events beginning after informed consent is obtained. Survey of other adverse events will be started after administration of the investigational product is started.
- d) Urine volume is measured for each void. A portion of the urine is collected, dispensed into a tube containing stabilizer, and stored frozen. The urine is forced to void at 24-hour intervals.

Group 2: Period I to IV

| · | Informed | Screening | | | Pe | rio d | I (B | : Do | sin | g 8 1 | 10U | rs af | te r b | igh- | fat r | ne a | l) | | | _ | | | Pe | riod | II ( | C: I | Dosi | ing 4 | 4 ho | urs : | afte | lov | -tat | me | al) | _ | | _ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day (time window) | consent | Day -30<br>to -2 | -1 | | | | | | | 1 | | | | | | | | | 2 | | | | | | | , | | 3 | _ | _ | | | | | | | 4 | |
| Time after dosing | | Visit | Admission | 8 h Pre-dose | Pre-dose | 0 | 5 m | 15m | 30 п | 45 m | 1 h | 1 1 30 ш | 2 h | 4. | 6 h | ч8 | 10 h | 12 h | 74 h | 36 h | 4 h Pre-dose | Pre-dose | 48 h | 0 | 5 m | 15 ш | 30 m | 45 m | 1.h | ш 0£ Ч І | 2 h | 4 h | 49 | 8h | 10 h | 12 h | 24 h | 36 h |
| Written informed consent | х | | | | | | | I | | | | | $\Box$ | | | | 1 | $\Box$ | I | $\Box$ | | | | Ľ | $\Box$ | | | | | | | $\Box$ | | | Ц | コ | | _ |
| Subject characteristics | | X | | | L., | | | | _ | _ | | _ | _ | | Ц. | $\perp$ | _ | _ | _ | _ | | L | ╙ | | Ш | | | | | $\Box$ | | _ | | | | _ | _ | |
| Eligibility assessment | | х | X | | Х | | | | | $\perp$ | | $\Box$ | | | _ | | _ | $\perp$ | _ | _ | | _ | | L | Ш | | | | _ | Ш | | _ | | | Ш | _ | _ | _ |
| Food (High Low Light)" | | | | High | | | | | | | | | _ | | | | | | | | Low | _ | | | Ш | | | | | | | _ | _ | | Ш | _ | _ | |
| Dosing of edaravone | | | _ | | _ | х | | _ | $\Box$ | | | | _ | _ | _ | _ | _ | _ | 4 | _ | | _ | <u> </u> | X | Ш | | ш | | | | | _ | _ | | Н | _ | _ | $\perp$ |
| Height, weight, BMI <sup>b)</sup> | | X | x | | | | | | | | | | | | | | | | | | | | | _ | | | | | | | | | _ | | Ш | | | |
| Physical examination | | х | x | | х | | П | | $\Box$ | | X | | | | | | | | x | | | X | | _ | | | | | Х | | | _1 | | | Ш | | X | _ |
| Vital signs | | х | X | | Х | | | | | | х | | | | | | | | ΧŢ | | | X | | $\perp$ | Ш | | | | Х | | | | _ | | Ш | | X | |
| 12-lead ECG | | X | х | | Х | | П | | | | Х | | | | | | $\perp$ | | x | | | X | l | L | | | | | х | L | | _ | _ | | Ш | | x | |
| Laboraty tests | | x | X | | Г | | $\Box$ | | | | | | | | $\perp$ | | | | _ | _ | | | | _ | | | Ш | | _ | Ш | | | _ | | Ш | $\perp$ | | |
| Serological tests | T | X | | | | | | | | | | | | | | _ | _ | $\perp$ | _ | _ | | $\perp$ | L. | ᆫ | | | | | | L., | | _ | _ | | Ш | _ | | _ |
| Drug/alcohol abuse screening | i | X | | | | | | | | | | | | _ | $\perp$ | _ | _1 | | _ | _ | | _ | | ┖ | | _ | | Ш | | | | | _ | | Ш | | | _ |
| Pregnancy test in female | | х | X | | | | | | | $\Box$ | | | | | | $_{\perp}$ | | $\perp$ | _ | _ | | <u>L</u> | ╙ | <u> </u> | Ш | | _ | | <u> </u> | | | | | Ш | Ш | $\sqcup$ | $\perp$ | _ |
| Adverse events () | <b>│</b> | ļ | Ε | | ⊢ | - | $\exists$ | $\exists$ | | | | - | - | $\pm$ | $\pm$ | $\pm$ | _ | $\pm$ | _ | ᆿ | | | 上 | | | | | | | | | | | | | = | | _ |
| Concomitant medications | | < | Н | | Е | F | $\exists$ | $\exists$ | | - | | | $\exists$ | 1 | 1 | - | -7 | $\exists$ | ∃ | = | | | Ė | | | | | | ⊏ | | | | = | | | = | | = |
| Blood sampling for edarayone | | | | | Х | | X | X | Х | X | Х | X | X | x | х | x | X | X : | Х | х | | | X | _ | X | X | Х | X | X | X | х | X | X | х | X | X | х | X |
| Urine sampling for edarayoned) | | | Т | | <b>\</b> | П | == | -7 | _ | $\neg \exists$ | L | = | $\pm$ | - | -Ŧ | ⊣ | - 7 | -T | $\dashv$ | $\neg$ | _ | - | ->< | - | Н | $\vdash$ | $\vdash$ | $\vdash$ | ┢ | Н | ├- | $\dashv$ | - | $\vdash$ | | _ | _ | _ |

| | | | | Pe | riod | Ш | (D: : | Dos | ing | 2 ho | urs | afte | r lig | ht n | neal | ) | | | | | | | Per | iod | IV ( | A: I | Dosi | ing 1 | ande | er fa | stec | l co | ndit | ion) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day (time window) | | | | | | | | | 5 | | | | | | | | | 6 | ; | | | | | | | | 7 | | | | | | | | 8 | 3 | 9 |
| Time after dosing | Before meals | 2 h Pre-dose | Pre-dose | 46 h | 0 | 5 m | 15 m | 30 m | 45 m | 1 h | 1 h 30 m | 2 h | 4 b | 6 h | 8h | 10 h | 12 h | 24 h | 36 h | Pre-dose | 48 h | 0 | 5 m | 15 m | 30 ш | 45 m | 116 | 1 h 30 m | 2 h | 4 h | 6 h | 8h | 10 h | 12 h | 24 h | 36 h | Discharge/48 h |
| Written informed consent | Ĺ | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | $\Box$ |
| Subject characteristics | | | | L | | | | | | | | | | _ | | L | _ | | | | | Ш | | | | | | <u>L</u> | | | <u> </u> | _ | ╙ | Ļ | 느 | ш | Ш |
| Eligibility assessment | | | | | | | _ | | | L | | 乚 | | | | 乚 | _ | | | | | Ш | | | | | | _ | | _ | _ | | L | _ | 辶 | ш | Ш |
| Food (High Low Light)*) | | Light | 1 | | | | | | | | | | | | | | | | L | | | | | | | Ш | | L., | | | L | | | 乚 | ㄴ | Ш | Ш |
| Dosing of edaravone | | | | | X | | | | | | | _ | | $oxed{oxed}$ | ᆫ | | _ | | _ | | | X | | | | | | 匚 | _ | ┖ | | | | ╙ | ₽ | L | Ш |
| Height,weight,BMIb) | | | П | Γ | | | | | | l | | | | | | _ | | | | | | | | | Ш | | | | | | | | <u> </u> | 上 | | 上 | Ш |
| Physical examination | Т | | X | | | | | | | X | Г | | | | | | | X | _ | Х | | | | | | | Х | L | | | _ | | L | | X | | х |
| Vital signs | Т | | X | | | | Г | | | X | | | | | | | | X | | Х | | | | | L | | Х | | | | _ | | _ | _ | X | | X |
| 12-lead ECG | | | X | П | | | | | | X | | | | | | | | X | | Х | | | | | | | X | | | | | | L | | X | 丄 | X |
| Laboraty tests | X | | Ī | П | | | | | | | | | | | | | | L | | | | | | | | | | | | | | <u> </u> | <u> </u> | ┖ | 上 | _ | X |
| Serological tests | | | | | | | | | | | | | | | | | | | | | | | | <u> </u> | <u> </u> | Ш | L | <u> </u> | 辶 | <u> </u> | | ┖ | <u> </u> | $\perp$ | L. | 辶 | Ш |
| Drug/alcohol abuse screening | | | | | | | | | | | | | 匚 | | Ĺ | $\perp$ | L | 乚 | | ᆫ | | | | L_ | 匚 | Ш | L. | <u> </u> | ╙ | <u> </u> | ╙ | $\perp$ | <u> </u> | ┖ | <b>Ļ</b> | ╙ | Ш |
| Pregnancy test in female | | | | L | L | | | | | | | | _ | | L | | | L | | | | | | ᆫ | <u> </u> | $oxed{oxed}$ | <u> </u> | <u> </u> | $\vdash$ | ┡ | <u> </u> | L | _ | $\perp$ | 上 | 丄 | Ш |
| Adverse events | ⇤ | ΕΞ | E | E | F | | | | | E | | E | $\vdash$ | | ╘ | | H | | | | | | | | - | | | | | = | ⇇ | | | E | 二 | 二 | ightharpoonup |
| Concomitant medications | ₩ | | E | Е | E | Е | | Ε | ╁ | E | H | E | Ē | E | ΙΞ | | | | | | | | | | ⊨ | | | | | | | | = | | Ħ | = | ď |
| Blood sampling for edaravone | | | | X | | X | Х | X | X | Х | X | X | X | X | X | X | X | X | X | | X | | х | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Urine sampling for edarayoned) | <b>(</b> | <del>-</del> | Ŧ | 1 | ŧ≂ | F | F | F | H | H | ⊢ | ⊦− | | 1 | +- | ╁ | $\vdash$ | ┼ | | - | $\times$ | 1 | $\vdash$ | Ι- | | <u> </u> | _ | | $\vdash$ | Η. | | $\vdash$ | $\vdash$ | t | 士 | 二 | $\rightarrow$ |

- a) High: High-fat meal, Low: Low-fat meal, Light: Light meal
- a) Height will be measured at screening only. Body weight will be measured at screening, admission, and end-of-study assessments. BMI will be calculated at screening and admission assessment.
- b) Assess serious adverse events beginning after informed consent is obtained. Survey of other adverse events will be started after administration of the investigational product is started.
- c) Urine volume is measured for each void. A portion of the urine is collected, dispensed into a tube containing stabilizer, and stored frozen. The urine is forced to void at 24-hour intervals.

Group 3: Period I to IV

| | | Screening | | ī | | erio | 41 | (C: 1 | Dosi | ing 4 | مدا | 115 | đer | low- | Set o | e al | ) | | П | | | P | erio | đΠ | D: | Dos | ing | 2 h | 1113 | a de | гlig | ht s | | 0 | _ | _ | 1 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day (time window) | Informed<br>consent | Day -30<br>to -2 | -1 | | | | _ | | | 1 | | | | | | | | 2 | | | | | | | | ` . | 3 | | | | | _ | | _ | | 4 | |
| Time after dosing | | Vait | Admission | 4 h Pre-dose | Pre-dose | 0 | | # 05 | 11 P. | H C+ | - 04.4. | 1 a 30 m | 4 | 49 | æ | 10 h | 12 b | 24 P | 36 h | 2 h Pre-dose | Pre-dose | 49 P | 0 | # S | 15m | 30 m | 45 m | 1.b | 1 h 30 m | 2 h | ₽<br>₽ | 6 h | 48 | 10 h | 13 h | 24 h | 4 82 |
| Written informed consent | X | | | | П | J | Ι | Т | Τ | Ι | Ι | | П | Ϊ | | | | | | | | П | | | | | | | | | _ | 4 | _ | 4 | _ | 4 | 4 |
| Subject characteristics | | X | | | | | | | _ | | L | | | | | | | | | | | Ц | Ц | Ц | _ | _ | _ | | _ | | _ | _ | _ | 4 | 4 | 4 | 4 |
| Eligibility assessment | | X | X | | X | | $\perp$ | П | | I | 1 | | | | | Ш | | | _ | | ш | Ц | Ш | | _ | _ | Ц | | | | _ | 4 | _ | _ | 4 | 4 | 4 |
| Food (High: Low: Light) <sup>a)</sup> | | | | Low | | | _ | | | l | 1 | | $\perp$ | | | | | | | Light | | Ш | | | | _ | _ | Ш | | _ | _ | _ | _ | _ | _ | 4 | 4 |
| Desing of educations | | | | | | X | I | Ι | I | $\perp$ | L | | | | | | | | | | L | Ш | X | | _ | | Ц | | | _ | Ц | _ | _ | _ | 4 | 4 | 4 |
| Height weight BMI <sup>h)</sup> | | X | X | | П | Т. | Ι | Т | Т | Т | Ι. | | | | | | | | | | | Ш | | | | | | | | | Ш | _ | _ | | _ | _ | 4 |
| Physical examination | | X | x | | X | | Ι | Т | Т | 72 | <u> </u> | $\perp$ | | | Ü | | | X | $\Box$ | | X | | | | | | Ц | X | | | Ц | _ | | _ | _ | X | 4 |
| Vital signs | | X | X | | X | 1. | Ι | | Ι | 7 | <u> </u> | $\perp$ | | | | | | X | | | X | L | | | | | Ц | X | | | Ц | _ | _ | _ | | X. | 4 |
| 12-lead ECG | | X | X | | X | Ι. | $\mathbf{I}$ | | | 7 | ζ. | | | | | | | X | $\Box$ | | X | Ш | Ш | | _ | | Ц | X | | | Ц | _ | _ | | 4 | X | 4 |
| Laboraty tests | | X | X | | $\Box$ | $\perp$ | Ι | | Ι | | Ι | Т | Г | $\Box$ | | | | $\Box$ | _ | | 匚 | $\sqcup$ | L | Ц | _ | | Ц | Ш | | _ | Ц | _ | Ц | Н | 4 | 4 | 4 |
| Serological tests | | X | L | | | | $\perp$ | | $\perp$ | $\perp$ | 1 | ┸ | ┸ | L | | Ш | Ш | Ц | | | ᆫ | L | _ | Ш | _ | | Ш | Щ | | | Ц | _ | Ц | Н | 4 | 4 | 4 |
| Drug/alcohol abuse screening | | X | | | | $\Box$ | Ι | | | $\perp$ | _ | ഥ | | L | | | Ш | Ц | | | L | $oldsymbol{\square}$ | | Ш | _ | | Ш | | | | Ц | | $\perp$ | Ш | 4 | 4 | 4 |
| Pregnancy test in female | | X | X | | | | | | | | 1 | ┸ | | | | Ш | Ш | Ц | _ | | ㄴ | ┖ | ш | Щ | _ | | Ш | Щ | Ц | Ц | Ц | _ | Н | Н | 4 | 4 | 4 |
| Adverse events | | | F | | $\Box$ | - E | $\pm$ | - | 1 | £ | £ | + | | | | Ш | | | | | | ㅂ | | $\exists$ | | | | | | | $\blacksquare$ | = | | Ħ | # | # | # |
| Concomitant medications | | | - | | Н | $-\mathbf{E}$ | Ε | H | Ŧ | Ŧ | 1 | £ | Ε | Ε | П | П | Н | $\exists$ | = | | | ㅂ | | Ħ | | | | | | | | = | | Ħ | # | ⇉ | # |
| Blood sampling for educatone | | | | | X | - 12 | r [ | X : | X 3 | X 2 | K [ | X X | X | X | X | X | X | X | X | | 上 | X | ட | X | x | X | X | X | X | X | X | I | X | X | X | 즤 | X. |
| Urine sampling for eduratione <sup>d)</sup> | | | Γ | | $\leftarrow$ | $\pm$ | - | | F | Ŧ | Ŧ | E | +- | +- | Ш | I | Н | $\Box$ | _ | | Ë | <b>&gt;</b> | $\vdash$ | П | $\dashv$ | | Н | Ш | - | - | ш | ⊒ | | | <u> </u> | # | # |

| | | _ | P | e rio | d 11 | I (A | : De | sin | ; w | der | fas | te d | COD | ditio | n) | _ | | Ĺ | | F | eric | dΓ | V (B | : De | sing | 8 1 | bour | 3 af | ter | igh | - Eut | me s | <u>5</u> | _ | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day (time window) | Г | | | | | | | 5 | | | | | | | | Γ | 6 | | | | | | | | 7 | | | | | | | | | 8 | 1 | 9 |
| Time after dosing | Pre-dose | 48 h | • | 5 28 | 15m | 30 m | 45 m | 1 1 | 1 h 30 m | 2 P | 4 | 9 | 48 | 101 | 12.8 | 24 % | 36 h | 8 h Pre-dose | Pre-dose | 48 b | 0 | S m | 15= | 30 ш | 45 m | 116 | 1 h 30 m | 2 h | 4.14 | <b>4</b> 9 | 8h | 10 h | 12 h | 24 b | 36 № | Discharge/48 h |
| Written informed consent | | | Т | | | | | | | | | t | t | Ĺ | Ĺ | | | | | | | | | | | | | | | | | | П | | | Ξ |
| Subject characteristics | | | Г | | | | | | | | L | | | L | | Ш | | | 1_ | ட | Ш | ட | Ш | $\Box$ | | ┖ | $oxed{oxed}$ | ᆫ | L | _ | | | L. | | ш | $\vdash$ |
| Eligibility assessment | | | | | | | | | L | <u>L</u> | L | | | _ | 上 | L | 上 | | <u> </u> | L | | oxdot | ᆫ | Ш | | | | ᆫ | _ | ╙ | _ | | L | _ | ш | _ |
| Food (High- Low- Light) | | | | | | | | | | | <u> </u> | | | L | | 1_ | | High | | | | | L | | | | | L | ட | _ | | | Ш | Ш | Ш | _ |
| Dosing of eduratione | Т | | Z | Γ | | | | Г | | | | Г | Г | | | L | | | | | X | | | | | | | L | ட | _ | _ | ┖ | Ш | Ш | Ш | _ |
| Height, weight, BMI <sup>b)</sup> | Т | П | Г | Г | | | | | | | | | Г | | | L | | | | <u>L</u> | | | | | | | | | 乚 | L | | | Ц | Ш | Ш | L |
| Physical examination | X | Т | Г | П | | П | | X | Г | Ι | Ι | Г | Т | Т | Τ. | X | | | X | | | | | | | X | | | L | | | | | X | Ш | X |
| Vital signs | X | | Г | | | | | Z | | | | | Г | | | Z | | | Z | L_ | <u> </u> | | | | | Z | | L | ட | _ | ᆫ | L | Ц | Z | Ш | X |
| 12-lead ECG | Z | 1 | Г | П | | | | X | | | | | Т | | | Z | | | Z | | | | | | | X | | L | ட | _ | ᆫ | L | Ш | Z | Ш | Z |
| Laboraty tests | X | | Γ | | | L | | | | | L | | | I | | L | L | | | | | <u> </u> | L | Ш | Ц | | | L | ᆫ | L | ᆫ | ╙ | Ш | $oxed{oxed}$ | Ш | Z |
| Serological tests | | | | $\Box$ | | | | | | | L | | Г | L | $\Box$ | L | $\Box$ | | ┖ | L | 匚 | 匚 | 匚 | oxdot | | | Ļ | L | L_ | <u> </u> | <u> </u> | <u> </u> | L | L | Ш | <u> </u> |
| Drug/alcohol abuse screening | | L | | | L | | 1_ | | | L | L | | L | | $\perp$ | $\perp$ | 上 | | 1 | <u> </u> | ┖ | 辶 | _ | L. | L. | ᆫ | <u> </u> | ┖ | ļ | ļ_ | _ | $\vdash$ | ᆫ | | Ш | L |
| Pregnancy test in female | | | | | L | L | | L | | | ┖ | L | | ┸ | ┸ | $\perp$ | 上 | | 1 | 乚 | 乚 | 乚 | 上 | ᆫ | | ╙ | ╙ | ᆫ | L | ᆫ | _ | <u> </u> | L | | ╙ | L |
| Adverse events | Е | F | F | F | Е | E | Н | | - | E | <del>-</del> | Ε | £ | $\pm$ | £ | $\pm$ | $\pm$ | ┢┈ | $\pm$ | <u>t</u> | | $\vdash$ | | | | | | ᆫ | 上 | | | ᆮ | | | | ₽ |
| Concomitant medications | E | Ŧ | Е | Н | Е | Е | Е | Е | E | Ŧ | Е | Ε | Ε | Ε | Ε | Ε | Е | | Η | ╁ | E | E | Ē | | | | | Ē | | | | | | = | | ightharpoonup |
| Blood sampling for edaratione | Z | Z | | X | Z | X | X | X | Z | Z | Z | Z | 7 | . 2 | 7 | z | Z | | $oxed{\Box}$ | Z | L | Z | X | Z | X | Z | X | X | X | X | X | X | Z | Z | Z | X |
| Urine sampling for edarayone <sup>d)</sup> | F | × | ļ | ⊢ | F | ₽ | +- | F | ⊢ | + | ┰ | + | ┰ | ┰ | + | +- | + | | + | <del>∤&gt;</del> ∙ | 1 | <del> </del> | + | <del> </del> | $\vdash$ | | | <u> </u> | | | <del></del> | _ | | <u>t </u> | $\vdash$ | ⇄ |

- a) High: High-fat meal, Low: Low-fat meal, Light: Light meal
- a) Height will be measured at screening only. Body weight will be measured at screening, admission, and end-of-study assessments. BMI will be calculated at screening and admission assessment.
- b) Assess serious adverse events beginning after informed consent is obtained. Survey of other adverse events will be started after administration of the investigational product is started.
- c) Urine volume is measured for each void. A portion of the urine is collected, dispensed into a tube containing stabilizer, and stored frozen. The urine is forced to void at 24-hour intervals.

Group 4: Period I to IV

| * * | Informed | Screening | | | Pe | ETÍO | ш | D: | Dosi | ng 2 | bot | ETS 2 | ner. | طها | i se | al) | | | | _ | | Pe | rio | П | (A: | Des | шg | | er 6 | sted | £01 | ناته | ) <u> </u> | ·- | _ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day (time window) | consent | Day -30<br>to -2 | -1 | | | | | | | 1 | | | | | | | | 1 | 2 | | | | | | _ | | 3 | | _ | | _ | | _ | L | 4 |
| Time after dosing | | Visit | Adm terion | 2 h Pre-dose | Pre-dose | 0 | 五 | 15 m | 30ж | 458 | - 01.4. | E PER I | 2 14 | <b>49</b> | <b>1</b> 8 | 101 | 12 h | 4 77 | 36 h | Pre-dose | 48 P | ٥ | 20.0 | 18 | 30 m | 45m | 4 | 1 h 30 m | 2 P | 44 | 5 | 40. | 121 | 24.6 | 1 1 |
| Written informed consent | X | | | | | | $\Box$ | $\Box$ | $\Box$ | I | Į | I | T | T | Ŧ | Ţ | Г | | | Ĺ | $\Box$ | 7 | 7 | 4 | 4 | $\dashv$ | Ц | $\dashv$ | 4 | $\bot$ | 4 | 4 | ╀ | ╀ | Ŧ |
| Subject characteristics | Ľ | X | L | | | | | _ | _ | _ | _ | _ | ㅗ | _ | ٠. | _ | ┺ | Ц. | ш | | _ | 4 | 4 | 4 | 4 | 4 | _ | _ | 4 | + | 4 | + | - | ╄ | + |
| Eligibility assessment | | X | X | | X | | | _ | | ┸ | ┸ | ┙ | | ┸ | 丄 | ┸ | L | <u> </u> | Ц | Ш | Ц | 4 | 4 | 4 | 4 | _ | _ | _ | 4 | Щ. | 4 | 4 | | ╄ | 4 |
| Food (High · Low Light) <sup>a)</sup> | | | Г | Light | | | | ┙ | | $\perp$ | ⊥ | ⊥ | 上 | 1 | | | | | L | | ш | _ | _ | _ | _ | _ | | Ш | Ц. | | _ | _ | ┸ | 1 | 4 |
| Dosing of educations | | | | | | X | | | | | | | | $\perp$ | I | L | | | | | | X | _ | _ | _ | _ | _ | Ш | 4 | _ | 4 | 4 | ┸ | 1 | 4 |
| Height,weight,BMI <sup>b)</sup> | | X | X | | П | | П | 7 | Т | Т | Т | Т | 1. | Ι | Т | | | L. | | | | | _1 | $\perp$ | | $\perp$ | | | ᆚ | $\bot$ | ı | $\perp$ | | L. | 丄 |
| Physical examination | † | X | x | | X | П | Т | ┪ | ┰ | 7 | X T | Т | Τ. | Ι | Т | Т | Г | X | | X | | | $\Box$ | П | | | X | | | $\perp$ | | | | 12 | |
| Vital signs | i – | X | X | | X | П | | П | Т | 7 | X [ | Т | Т. | Τ | Т | T | | X | | X | | | $\Box$ | | | | X | | | $\perp$ | | $\perp$ | L | 13 | |
| 12-lead ECG | 1 | X | Ī | | X | | П | ╗ | Т | 1: | xΤ | Т | Т | Т | Т | Т | Ι | X | | X | | | | | | | X | | $\perp$ | ユ | _ | | 1. | 12 | ٢. |
| Laboraty tests | | x | Ī | | П | $\neg$ | Т | ╗ | ┑ | T | Т | Т | | Т | Т | | Τ | | | | | | $\Box$ | | | | | | _ | 丄 | _ | | 1 | L | ┸ |
| Serological tests | | х | Г | | | | | | | | | $\Box$ | | | | | L | L_ | Ш | | | ┸ | _1 | | | | | | _ | _ | ┸ | _ | ┸ | ┸ | 4 |
| Drug/alcohol abuse screening | 1 | х | Г | | | | | | | Ι | Т | $\Box$ | П., | Ι | | L | Ц | | | | | | _ | _ | _ | | | | _ | _ | 4 | Ц. | ┸ | Ţ. | 4 |
| Pregnancy test in female | T | X | X | | | | I | Ι | | Ι | I | $\perp$ | | $\perp$ | | Г | Г | | | | Ц | _ | _ | _ | _ | _ | | Ц | _ | 4 | 4 | 1 | ┸ | 1 | 4 |
| Adverse events <sup>e)</sup> | <b></b> | | F | | H | $\blacksquare$ | $\exists$ | $\exists$ | $\exists$ | $\pm$ | 1 | 1 | | Ξ | Ė | $\pm$ | + | 上 | $\vdash$ | Н | | ⇉ | _ | | ╛ | ⇉ | | | _ | # | # | 1 | # | 1 | + |
| Concernitant medications | 1 | <del></del> | F | | | | $\exists$ | = | $\blacksquare$ | | = | Ŧ | Ŧ | Ξ | | - | $\pm$ | Ε | Н | Ш | Ī | Ŧ | $\exists$ | $\equiv$ | $\exists$ | $\exists$ | _ | | Ⅎ | # | 1 | Ŧ | 1 | 1 | + |
| Blood sampling for educatone | T | | Т | | x | | X | X | X | X : | X : | xΤ | XX | ( ) | C X | X | X | X | X | X | Х | _ | x | ΣŢ | X | X | X | X | ΧŢ | X : | X : | X 2 | | 13 | 4 |
| Tiring complime for adarwage <sup>(i)</sup> | | Ĭ . | Т | | ₩ | | $\dashv$ | 7 | $\dashv$ | 7 | 7 | =Ŧ | Ŧ | - | Ŧ | + | 1 | F | Ε- | | X | -Ŧ | -1 | 7 | - | | - | $\vdash$ | $\mathbf{I}$ | $\pm$ | - | $\pm$ | 1 | ± | + |

| | | | Per | iod l | W ( | B: I | Dosi | ng 8 | bo | ars. | s∄e | r b | igh | Set : | De x | J) | | | I | | _ | | Pe | riod | W | (C: | Dos | ing. | 4 L | ) WES | afte | r lo | r L | | 3) | _ | _ | = | コ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day (time window) | | | | | | | | 5 | | | | | | | | | | 6 | | | | | | | | | 7 | | | | | | | | | 1 | В | 9 | |
| Time after dosing | 8 h Pre-dose | Pre-dose | 48 h | 0 | 5 m | 15 m | 30 m | 45 = | 11 | 1 1 30 | 2 h | 7 | | | | | | 24 h | 36 h | 4 h Pre-dose | Pre-dose | 48 P | 0 | 5 m | 15 m | 30 88 | đã m | = | 1 h 30 m | 2.1 | 4.1 | 19 | 48 | 10 h | 121 | 24 h | 36 h | 46h | Discharge/48 h |
| Written informed consent | | | | | | | | | | | | | Ι | Ţ | T | | T | | ┒ | | | | | | | | Г | | | | | | | | | | | Ш | コ |
| Subject characteristics | | | | | | | | | | | L | L | L | $\perp$ | 1 | ┸ | ᆚ | | _ | | Ш | L | L | 辶 | ᆫ | ᆫ | ᆫ | ᄂ | ┖ | | 辶 | Ш | | | | ╙ | ┅ | <u> </u> | _ |
| Eligibility assessment | | | | | | | | | | | L. | L | L | ⊥ | ┸ | ┸ | ┸ | _ | _ | | 乚 | L | ᆫ | <u>L</u> | ┖ | ᆫ | ᆫ | L | ᆫ | | ᆫ | 上 | _ | | | L | ╙ | ш | _ |
| Food (High: Low: Light)*) | High | | | | | | | | | | | | | L | | - | | | | Low | | L | L | L | | L | | | 1_ | | | L | Ш | | ш | _ | ш | Ш | _ |
| Dosing of edaratone | | П | П | X | | | | | | | Γ | Г | Т | Ι | Т | 1 | Т | $\exists$ | | | | Ĺ | Z. | L | | | | | L | | | | Ш | | _ | Ш | ┖ | ш | _ |
| Height, weight, BλΠ <sup>b)</sup> | | П | | П | | | | | | Г | Г | Г | Т | Т | Т | Т | Т | Т | 7 | | Г | I | | | П | | | 1 | I _ | | | | | | | | L | Ш | |
| Physical examination | | Z | П | | | | Ξ | | Z | | T | Г | T | $\top$ | Т | T | 7 | X | 1 | | Z | | | | | | | X | | | | | | | ட | Z | | | X |
| Vital signs | | X | | | | | П | | X | Г | T | Г | Т | Т | Т | Т | | X | Т | | Z | Г | | | | | | X | | | | | | | ட | X | ட | Ш | X |
| 12-lead ECG | | X | П | | | | | | Z | | Г | Г | Т | Т | Т | Т | Т | $\overline{\mathbf{x}}$ | _ | | Z | Г | | | | | | Z | L | | | | | | ட | X | ட | Ш | X |
| Laboraty tests | | Z | П | П | | | | | | | Г | Γ | Τ | Т | Τ | Т | Т | $\Box$ | $\Box$ | | | | | 匚 | | | | | L | | 乚 | | | | ᆫ | ┖ | ᆫ | Ц | Z |
| Serological tests | | 1 | П | П | | | | | | | Г | Т | $\mathbf{I}$ | | | | | $\Box$ | | | | | L | L | L | L | 乚 | 上 | L | ┖ | ᆫ | 乚 | | | 匚 | ┖ | ᆫ | Ш | Ш |
| Drug/sicohol abuse screening | | 1 | П | П | | | | | | | Г | Ι. | Ι | | | | | | | | | | L | L | L | 上 | L | 上 | L | L | | 辶 | | _ | ட | ᆫ | ᆫ | Ш | |
| Pregnancy test in female | | 1 | | Γ | | | | | | | L | | $\perp$ | ⊥ | | | $\perp$ | | | | 匚 | | L | L | 上 | 乚 | 上 | 上 | L | 丄 | _ | <u> </u> | L | <u> </u> | ᆫ | ╙ | ┖ | Ш | المرا |
| Adverse events <sup>e)</sup> | k | F | | | _ | Н | Н | Н | - | $\vdash$ | ₽ | ₽ | Ŧ | $\pm$ | - | $\pm$ | - | $\exists$ | $\exists$ | | 1 | | Ė | | Ŀ | <u> </u> | ╁ | $\pm$ | | $\perp$ | _ | 上 | ᆮ | | | ╧ | ᆮ | ᆸ | ightharpoonup |
| Concountant medications | <b>K</b> | ⊨ | F | | - | Е | F | $\vdash$ | | - | F | Е | Ŧ | Ŧ | Ε | Ŧ | Ŧ | $\exists$ | $\exists$ | | E | Е | Е | | | | Е | Ŧ | Е | | - | E | | | | | 三 | | ᅼ |
| Blood sampling for edaratione | | | X | | X | X | Z | X | Z | X | Z | 3 | 3 | ς : | <b>X</b> | X | Z | Z | X | | | Z | | Z | Z | X | X | Z | Z | X | Z | X | X | X | X | Z | X | X | ш |
| Urine sampling for edarsyone <sup>4)</sup> | <b></b> | F | × | - | П | П | Е | Е | Е | | F | F | E | $\pm$ | $\pm$ | Ŧ | $\pm$ | - T | $\exists$ | | Ε | × | Ε | E | ⇇ | Ε | Ⴞ | E | 上 | 巨 | | Ė | ᆫ | | ᆂ | | 上 | ᆸ | ightharpoons |

- a) High: High-fat meal, Low: Low-fat meal, Light: Light meal
- a) Height will be measured at screening only. Body weight will be measured at screening, admission, and end-ofstudy assessments. BMI will be calculated at screening and admission assessment.
- b) Assess serious adverse events beginning after informed consent is obtained. Survey of other adverse events will be started after administration of the investigational product is started.
- c) Urine volume is measured for each void. A portion of the urine is collected, dispensed into a tube containing stabilizer, and stored frozen. The urine is forced to void at 24-hour intervals.

# All groups: Period V

| Day (time window) | | | | | | | | | I | e ric | d V | ,<br> | | | | | | | | End-of-study<br>assessment <sup>e)</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | X | | | | | | | | X+1 | | | | | | | | X- | +2 | X+3 | X+8 (±2) |
| Time after dosing | Admission | b) " h Pre-dose | Pre-dose | 0 | 5 m | 15 m | 30 m | 45 m | 1 h | 1 h 30 m | 2 h | 4 h | 6 h | 8h | 10 h | 12 h | 24 h | 36 h | Discharge/48 h <sup>9</sup> | Visit |
| Food *) | | X | | | | | | | | | | | | | | | | | | |
| Dosing of edaravone | | | | X | | | | | | | | L. | | | | | | | | |
| Weight | X | | | | | | L. | | | | | _ | | | | | <u> </u> | | | X |
| Physical examination | X | | X | | L | | | _ | X | | | | | <u>L</u> | | | X | | X | X |
| Vital signs | X | | X | | | | | | X | | | ļ | | | | <u> </u> | X | | X | X |
| 12-lead ECG | X | | X | | | | L_ | | X | | L. | _ | | | | | X | | X | X |
| Laboraty tests | X | | | | <u> </u> | | | | | <u> </u> | _ | | | | | | | L | X | X |
| Pregnancy test in female | <u> </u> | | | | | | | | | | | | _ | | | | | <u> </u> | | X |
| Adverse events c) | ← | | | | | | | | | | | | | | | | | | ightharpoons | |
| Concomitant medications | $\lor$ | E | | | | | | | | | | | | | | _ | | | > | |
| Blood sampling for edaravone | _ | | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Urine sampling for edaravone d) | | | <b>←</b> | | | | | | | | _ | <u> </u> | | | | | | | $\Rightarrow$ | |

- a) The diet menu in period V will be determined based on the PK data collected from period I to IV.
- b) The dosing time after a meal in period V will be determined based on the PK data collected from period I to IV.
- c) Assess serious adverse events beginning after informed consent is obtained. Survey of other adverse events will be started after administration of the investigational product is started.
- d) Urine volume is measured for each void. A portion of the urine is collected, dispensed into a tube containing stabilizer, and stored frozen. The urine is forced to void at 24-hour intervals.
- e) At the time of withdrawal, the same tests will be performed as those of the end-of-study assessment.
- f) In the F: Dosing 4 hours after light meal, tests/observations are conducted 46 hours after administration of the investigational product.

# 3.4. Sample Size and Power Considerations

Total of 16 subjects (4 subjects per group)

[Rationales for setting]

The target number of subjects was set on the assumption that it would allow obtaining results that will meet the study objectives although it is not based on statistical calculations.

# 4. PLANNED ANALYSIS

#### 4.1. Final Analysis

This SAP will be finalized before database lock. Final data analysis will be conducted after database lock.

#### 5. ANALYSIS POPULATIONS

PK analysis will be performed on the PK analysis set. Safety analysis will be performed on the safety analysis set (SAF). The definitions of the analysis sets are provided below. The detailed handling of subjects was determined by the sponsor, by the time of the data lock.

# (1) PK analysis set

The PK analysis set will consist of all subjects who received at least 1 dose of the investigational product and had evaluable PK data.

(2) Safety analysis set

The SAF will consist of all subjects who received at least 1 dose of the investigational product.

# 6. STATISTICAL CONSIDERATIONS

#### 6.1. Descriptive Statistics

#### (1) Non-PK related

Continuous data will be summarized descriptively using the number in the analysis set (N), the number of observations (n), mean, standard deviation (SD), median, minimum and maximum. Categorical data will be summarized using frequency counts and percentages. The denominator for the percentages will be the total number of subjects in the treatment group and analysis population being presented, unless otherwise specified.

# (2) PK related

Plasma concentrations will be summarized descriptively using N, n, mean, SD, median, minimum and maximum.

The plasma and urine PK parameters will be summarized descriptively using N, n, arithmetic mean, SD, median, CV%, range (minimum, maximum), geometric mean and geometric CV% CV% and Geometric CV% will be calculated as follows:

$$CV\% = \frac{\text{standard deviation}}{\text{arithmetic mean}} \times 100$$

Geometric CV% = 
$$\sqrt{[\exp(\sigma^2) - 1]} \times 100$$

where  $\sigma$  represents the standard deviation computed on the natural logarithmic transformed concentrations.

#### 6.2. Statistical Tests

Unless otherwise specified, all formal statistical tests of treatment effects will be done at two-sided significance level of 0.05. Point estimates will be accompanied with two-sided 95% CIs where applicable.

# 6.3. Data Review Meeting

Prior to database lock, a data review meeting (DRM) was conducted at November 26, 2019. Protocol deviation and handing of subjects and records, for analysis sets and evaluations, was confirmed during DRM.

No protocol deviation was observed during the study. As a results of DRM, all subject was included in SAF and PK analysis set.

The PK data handling was assessed during DRM. All PK data were considered valid and included in the calculation of PK parameters and in the summary tables and figures.

#### 7. DATA CONVENTIONS

#### 7.1. Analysis Variable Definitions

#### 7.1.1. Study Subjects

# 7.1.1.1. Demographic and Other Baseline Characteristics

#### (1) BMI

BMI will be recalculated using the formula below and reported to 1DP.

BMI  $(kg/m^2)$  = weight at Day -1 (kg) / {height at screening (m)}<sup>2</sup>

(2) Age at informed consent

Age (year) = year of informed consent – year of birth

Subtract 1 from the age (years) calculated above, if [Month of informed consent < Month of birth] or [Month of informed consent = Month of birth AND Day of informed consent < Day of birth].

#### 7.1.1.2. Medical History

Medical history will be coded according to the MedDRA version 22.0.

#### 7.1.1.3. Prior or Concomitant Medication

Medications will be coded according to the WHO Drug Global B3 Format March 1, 2019.

#### (1) Prior Medication

Prior medication is any medication that was stopped prior to the investigational product administration.

#### (2) Concomitant Medication

The investigator (or subinvestigator) will confirm whether each subject has used any medications (including commercially available drugs) other than the investigational product, between the start of investigational product administration and completion of the end-of-study assessment.

# 7.1.2. Safety Assessments

#### 7.1.2.1. Adverse Events

Adverse events will be coded according to the MedDRA version 22.0

(1) Adverse Events/ Serious Adverse Events (AEs/SAEs)

An AE/SAE is any untoward medical occurrence or unintended sign (including an abnormal laboratory finding), symptoms, and disease in a patient or subject who is administered a pharmaceutical product during safety assessment period, and which does not necessarily need to have a causal relationship with the treatment.

(2) Adverse Drug Reaction

A AE is considered "adverse drug reaction" if it has been assessed as having a "reasonable possibility" in relationship to the investigational product.

(3) Time to Adverse Events

Time to Adverse Events occurrence (days) = AE start date – date of first administration + 1

(4) Duration of Adverse Events

Duration of Adverse Events (days) = AE stop date – AE start date + 1

# (5) Period of Adverse Events

| | Se Events | | | |
|---|---|---|---|---|
| Visit in Group 1 | Visit in Group 2 | Visit in Group 3 | Visit in Group 4 | For TFLs |
| From on or after | From on or after | From on or after | From on or after | Fasted |
| administration | administration | administration | administration | |
| date/time in Day | date/time in Day | date/time in Day | date/time in Day | |
| 1 to before | 7 to before | 5 to before | 3 to before | |
| administration | administration | administration | administration | |
| date/time on in | date/time on in | date/time on in | date/time on in | |
| day 3 | day 23 | day 7 | day 5 | |
| From on or after | From on or after | From on or after | From on or after | 8 hours |
| administration | administration | administration | administration | after high- |
| date/time in Day | date/time in Day | date/time in Day | date/time in Day | fat meal |
| 3 to before | 1 to before | 7 to before | 5 to before | |
| administration | administration | administration | administration | |
| date/time on in | date/time on in | date/time on in | date/time on in | |
| day 5 | day 3 | day 23 | day 7 | |
| From on or after | From on or after | From on or after | From on or after | 4 hours |
| administration | administration | administration | administration | after low- |
| date/time in Day | date/time in Day | date/time in Day | date/time in Day | fat meal |
| 5 to before | 3 to before | 1 to before | 7 to before | |
| administration | administration | administration | administration | |
| date/time on in | date/time on in | date/time on in | date/time on in | |
| day 7 | day 5 | day 3 | day 23 | _ |
| From on or after | From on or after | From on or after | From on or after | 2 hours |
| administration | administration | administration | administration | after light |
| date/time in Day | date/time in Day | date/time in Day | date/time in Day | meal |
| 7 to before | 5 to before | 3 to before | 1 to before | |
| administration | administration | administration | administration | |
| date/time on in | date/time on in | date/time on in | date/time on in | |
| day 23 | day 7 | day 5 | day 3 | |
| From on or after | From on or after | From on or after | From on or after | 2 hours |
| administration | administration | administration | administration | after low- |
| date/time in Day | date/time in Day | date/time in Day | date/time in Day | fat meal |
| 23 to end of study | 23 to end of study | 23 to end of study | 23 to end of study | |
| assessment | assessment | assessment | assessment | |

# 7.1.2.2. Laboratory Tests

Values for out of pre-defined clinically relevant will have clinically relevant values flagged set (L=Lower than normal range, H=Higher than normal range or A=Abnormal).

#### 7.1.2.3. 12-Lead ECG

(1) Criteria for pre-defined limit

12-lead ECG:

- QTcF > 500msec
- 500 >= QTcF > 480msec
- $480 \ge QTcF \ge 450$ msec
- QTcF <= 450 msec
- Change from baseline in QTcF > 30 msec
- Change from baseline in QTcF > 60 msec

#### 7.1.3. Pharmacokinetics Evaluation

# 7.1.3.1. Plasma Concentration

For the calculation of the summary statistics, concentration values reported as below the limit of quantification (BLQ) will be set to 0.

#### 7.1.3.2. Pharmacokinetic Parameters

Below the limit of quantification

For the calculation of PK parameters, actual sampling time (in hours rounded to 3 DPs) relative to dosing should be used. Concentration below the limit of quantification (BLQ) will be imputed with a value of 0. For calculation of AUCs, missing data will be treated as if the respective sample never had been scheduled for the calculation by the linear-linear trapezoidal rule. For Ae, Ae% and CLr, geometric mean and geometric CV% will be calculated only when all the individual Ae, Ae% and CLr is greater than 0 in each sampling time point.

# 7.2. Analysis Visit Definitions

# (1) Non-PK related

The date of the first dose of investigational product is defined as Day 1.

Excepted for laboratory, baseline will be the last observed value of the parameter of interest prior to the first intake of investigational product by each treatment period (this includes unscheduled visits). For laboratory, baseline will be the last observed value of the parameter of interest prior to the first intake of investigational product (this includes unscheduled visits).

No analysis visit window will not be perfored for safety evaluation.

# (2) PK related

The allowable time window will be the following.

Plasma PK sampling

| Nominal Time Point | Window |
|---|---|
| Predose | Within 60 min before dosing |
| 0.083 h after dosing | Nominal time point ± 1 min |
| 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12 h | Nominal time point ± 5 min |
| after dosing | |
| 24, 36 h after dosing | Nominal time point $\pm$ 15 min |
| 48 h* after dosing | |
| *Following the dosing 4 hours after | |
| meals, blood sampling is conducted | |
| 46 h after dosing | |
| Blood sampling 46 h after dosing | [Period I, II, and III] 45~47 h after dosing |
| | and within 60 min before the dosing in |
| | the next period |
| | [Period IV and V] 45~47 h after dosing |
| Blood sampling 48 h after dosing | [Period I, II, and III] 47~50 h after dosing |
| | and within 60 min before the dosing in |
| | the next period |
| | [Period IV and V] 47~50 h after dosing |

Urine PK sampling

| Nominal Time Point | Window |
|-----------------------------------------|-----------------------------|
| Predose | Within 60 min before dosing |
| Voluntary Urine | _ |
| Forced micturition at 24 h after dosing | Nominal time point ± 30 min |

| Nominal Time Point | Window |
|---|---|
| Forced micturition at 48* hours post-dose | · |
| * Forced micturition at 46 h post-dose | |
| for subjects dosed 4 h after meals | |
| Forced micturition at 46 h after dosing | [Periods I, II, and III] 45~47 h after |
| | dosing and within 60 min before the |
| | dosing in the next period |
| | [Periods IV, V] 45-47 h post-dose |
| Forced micturition at 48 h after dosing | [Periods I, II, and III] 47~50 h after |
| | dosing and within 60 min before the |
| | dosing in the next period |
| | [Periods IV, V] 47~50 h post-dose |

# 7.3. Data Handling Convention for Missing Data

#### (1) Non-PK related

#### Adverse events:

If severity or relationship is found to be missing the most severe occurrence will be imputed for the summary of interest.

# Other safety:

For safety summaries, only observed data will be used. Unless otherwise specified, missing safety data will not be imputed.

# (2) PK related

For PK summaries, only observed data will be used. Missing PK data will not be imputed. When calculating Ae and Ae%, missing PK data will be imputed to 0.

# 8. STATISTICAL METHODOLOGY

# 8.1. Study Subjects

# 8.1.1. Subject Disposition

Subject disposition will be summarized on the SAF and listed on the enrolled subjects.

# 8.1.2. Analysis Populations

Analysis populations including the inclusion and exclusion criteria deviation at screening will be summarized and listed on the all enrolled subjects.

# 8.1.3. Administration of Investigational Product

Administration data will be summarized and listed on the SAF.

# 8.1.4. Demographic and Other Baseline Characteristics

The following demographic and other baseline characteristics will be used.

| | category | descriptive |
|---|---|---|
| Sex | Male, Female | |
| Age at informed consent(years) | | Yes |
| Height(cm) | | Yes |
| Weight(kg) | | Yes |
| BMI(kg/m <sup>2</sup> ) | | Yes |
| Race | Japanese | |
| Medical<br>History | No, Yes | |
| Complication | No (if status ofmedical history is 'Ongoing'), Yes (if otherwise) | |
| Concomitant<br>Medication | No, Yes | |
| Allergic<br>History<br>(including drug<br>allergies) | No, Yes | |
| Drinking Status | No (if 'Never'), Yes (if otherwise) | |
| Smoking Status | No (if 'Never'), Yes (if otherwise) | |

Demographic and other baseline characteristics will be summarized and listed on the SAF.

# 8.1.5. Medical History and Allergic History

Medical history and allergic history will be listed on the SAF.

# 8.1.6. Prior or Concomitant Medications

Prior and concomitant medication will be listed on the SAF.

# 8.2. Efficacy Assessments

N/A

# 8.3. Safety Assessments

Safety assessments will be made on the SAF population.

#### 8.3.1. Adverse Events

Overall summary for the following will be conducted by treatment.

- Subjects with at least one AE
- Subjects with at least one adverse drug reaction
- Subjects with at least one SAE
- Subjects with at least one serious adverse drug reaction
- Subjects with at least one AE leading to discontinuation of investigational product
- Subjects with AE leading to death

The following summaries also will be conducted by treatment.

- AEs by SOC and PT
- Adverse drug reactions by SOC and PT
- AEs by SOC, PT and severity

Each of the summaries will be done at the subject level - multiple occurrences of the same event within a subject will be counted once in the summaries by SOC and PT; multiple occurrences of the same event within a subject will be counted once in the maximum severity category (severe > moderate > mild) and/or maximum drug relationship category (reasonable possibility/no reasonable possibility) and/or the earliest duration.

All AEs will be listed.

# 8.3.2. Laboratory Tests

Absolute values and changes from baseline, except for urinalysis will be summarized descriptively by group and scheduled visit.

For urinalysis, number and percentage will be presented. Shift tables will present the changes in clinically relevant categories from baseline to each scheduled post-baseline visit by group and scheduled visit.

Below in a list of the laboratory test.

| Laboratory Test | Parameters |
|---|---|
| Hematology | Hemoglobin, hematocrit, red blood cell count, white blood cell count, platelet count, MCH, MCHC, MCV, differential white blood count |
| Biochemistry | Na, K, Cl, Ca, inorganic phosphorus, urea nitrogen, creatinine, uric acid, total bilirubin, direct bilirubin, ALT, AST, γ-GTP, ALP, LDH, CK, amylase, total cholesterol, triglycerides, LDL-C, HDL-C, total protein, albumin, glucose |
| Coagulation test | Prothrombin time, activated partial thromboplastin time |
| Urinalysis | Qualitative tests (pH, specific gravity, protein, glucose, occult |
| | blood, urobilinogen, bilirubin, ketones), sediment(listing only) |

All data including clinically relevant flagged will be listed. Any BLQ data will be treated as 0 in summary statistics.

# 8.3.3. Vital Signs

Absolute values and changes from baseline will be summarized for the following parameters by treatment and scheduled time point.

- Systolic Blood Pressure (mmHg)
- Diastolic Blood Pressure (mmHg)
- Pulse Rate (bpm)
- Body Temperature(°C)

All data will be listed.

#### 8.3.4. 12-Lead ECGs

Absolute values and changes from baseline will be summarized for the following parameters by treatment and scheduled time point.

- Heart Rate (beats/min)
- PR (msec)
- RR (msec)
- QRS (msec)
- QT (msec)
- QTcF (msec)

The percentage of subjects with 12-lead ECG values outside pre-defined limit will be summarized by treatment and scheduled time point.

All data (including overall evaluation) will be listed.

# 8.3.5. Physical Examinations

Physical examination will be listed.

#### 8.4. Pharmacokinetics Evaluation

Summaries of concentrations, PK parameters and statistical analysis for unchanged edaravone, sulfate conjugate, and glucuronide conjugate will be performed using data from subjects whose PK data will be available in at least one treatment.

# 8.4.1. Concentrations and Pharmacokinetic Parameters for unchanged edaravone, sulfate conjugate, and glucuronide conjugate

Plasma unchanged edaravone, sulfate conjugate, and glucuronide conjugate concentrations will be summarized at each nominal sampling point for each treatment. All plasma concentrations will also be listed.

For each treatment, individual plasma concentrations vs. actual time for unchanged edaravone, sulfate conjugate, and glucuronide conjugate will be plotted on both linear/linear and log/linear scales. Mean plasma concentrations vs. nominal time curves will be plotted on both linear/linear (+SD) and log/linear scales overlaid by each treatment.

The PK parameters listed in Section 2.2.2 will be calculated for each subject using non-compartmental model. The PK parameters will be listed and summarized by each treatment. The PK parameters listed as other PK parameters will not be summarized. The urinary pharmacokinetic parameters will be listed and summarized for each treatment. The urinary pharmacokinetic parameters at pre-dose will not be summarized.

# 8.4.2. Analysis of Food Effect

The parameters  $C_{max}$ ,  $AUC_{0-\infty}$ ,  $AUC_{0-24}$ , and  $AUC_{0-t}$  of unchanged edaravone will be log transformed prior to statistical analysis. For period 1 to 4, the analysis will be by analysis of variance (ANOVA) taking account of meal conditions. Factors accounting for the following sources of variation: sequence, subjects nested in sequences, periods, and meal conditions. For subjects having each value with fasted and period 5, the analysis will be by ANOVA taking account of meal conditions. Factors accounting for the following sources of variation: sequence, subjects nested in sequences, and meal conditions. Difference in least square (LS) means and corresponding 90% CI will be back transformed to obtain the estimate and CI of geometric mean ratio of each meal conodition to fasted. As reference, the same analysis will also be on sulfate conjugate and glucuronide conjugate.

For  $C_{max}$ , and  $AUC_{0-\infty}$  spagnetti plots will be produced showing individual differences between fasted condition and each meal condition.

# 9. DATA PRESENTATION CONVENTIONS

# 9.1. Number of Digits to Report

# (1) Non-PK related

| Statistic | Specification | Apply to |
|---|---|---|
| Minimum, Maximum | Same number of DPs as the data provided in the datasets | All original (i.e. non-derived) |
| | see section 7.3 | All derived data |
| Mean, Median, SD, SE,<br>Confidence intervals | One more DP than above | All |
| Percentages*1 | 1 DP | All |

<sup>\*1</sup> Percentages: use 1 place beyond the decimal point, except for the following cases:

If the percentage is equal to 0, then leave blank, do not use (0)

If the percentage is equal to 100, then use "(100)" without a decimal

# (2) PK Plasma Concentration

| Statistic | Specification |
|--------------------|---------------------------------------------------|
| Individual value | With the number of DPs to which they are reported |
| Mean, SD, Minimum, | Same number of DPs as the individual value |
| Median, Maximum | |

# (3) PK Parameters

# Plasma PK Parameters

| Statistic | Specification |
|---|---|
| Individual value | C <sub>max</sub> : same number of DPs as the plasma concentration |
| | t <sub>max</sub> *: 2 DPs |
| | Kel: 4 DPs |
| | Other parameters to be summarized: number of DPs |
| | which the number of significant digits of a minimum |
| | parameter is three |
| | AUC% <sub>ex</sub> : 2 DPs |
| | Adjusted R <sup>2</sup> : 2 DPs |
| | Number of Kel points: 0 DP |
| | Lower and Upper limited of Kel: 2 DPs |
| Mean, SD, Minimum, | Same number of DPs as the individual values |
| Maximum, Median, | |
| Geometric mean | |
| CV%, Geometric CV% | 1 DP |
| Ratios | 3 DPs |

<sup>\*:</sup> t<sub>max</sub> will be expressed basically in terms of median and range

# Urine PK Parameters

| Statistic | Specification |
|------------------|----------------|
| Individual value | Ae, Ae%: 3 DPs |

| | CLr: number of DPs which the number of significant |
|--------------------|----------------------------------------------------|
| | digits of a minimum parameter is three |
| Mean, SD, Minimum, | For Unchanged Edaravone: 3 DPs |
| Maximum, Median, | For Sulfate Conjugate: 2 DPs |
| Geometric mean | For Glucuronide Conjugate: 1 DP |
| | For Sum of Unchanged Edaravone and Metabolites: |
| | 1 DP |
| CV%, Geometric CV% | 1 DP |

# 9.2. Treatments to Report

| Treatment | For TFLs |
|------------------------------------|-----------------------------|
| Dosing under fasted condition | Fasted |
| Dosing 8 hours after high-fat meal | 8 hours after high-fat meal |
| Dosing 4 hours after low-fat meal | 4 hours after low-fat meal |
| Dosing 2 hours after ligh meal | 2 hours after light meal |
| Dosing 2 hours after low-fat meal | 2 hours after low-fat meal |

# 9.3. Analysis Visits to Report

# (1) Non-PK related

| Analysis Visit | Analysis Time Point | Apply to | | |
|---|---|---|---|---|
| | | Laboratory | Vital Signs | 12-Lead ECGs |
| | | Tests | | |
| Screening | | X | X | X |
| Day -1 | | X (baseline) | X | X |
| Day 1 | Pre-dose | | X (baseline) | X (baseline) |
| Day 1 | 1 hour | | X | X |
| Day 2 | 24 hours | | X | X |
| Day 3 | Pre-dose | | X (baseline) | X (baseline) |
| Day 3 | 1 hour | | X | X |
| Day 4 | 24 hours | | X | X |
| Day 5 | Pre-dose | X | X (baseline) | X (baseline) |
| Day 5 | 1 hour | | X | X |
| Day 6 | 24 hours | | X | X |
| Day 7 | Pre-dose | | X (baseline) | X (baseline) |
| Day 7 | 1 hour | | X | X |
| Day 8 | 24 hours | | X | X |
| Day 9 | 46 hours | X | X | X |
| Day 23 | | X | X | X |
| Day 24 | Pre-dose | | X (baseline) | X (baseline) |
| Day 24 | 1 hour | | X | X |
| Day 25 | 24 hours | | X | X |
| Day 26 | 48 hours | X | X | X |
| Follow up | | X | X | X |

Screening, unscheduled visits, retests (same visit number assigned) will not be displayed in byvisit summary tables, but will be included in the data listings.

# 10. CHANGE FROM THE PROTOCOL

There are currently no changes to analysis from protocol.

# 11. SOFTWARE

All statistical analyses will be performed using SAS version 9.4 or higher. The PK parameters will be calculated using WinNonlin® software (version 6.3 or later).

# 12. REFERENCES

N/A

# Appendix 1 Pharmacokinetic Parameter Calculations

- Actual blood sampling times will be used in the calculation of pharmacokinetic parameters
- All concentrations below the LLOQ will be set at zero for pharmacokinetic calculations
- When Kel is missing (or cannot be determined), t<sub>1/2</sub>, AUC<sub>0-∞</sub>, AUC<sub>0-∞</sub>, AUC<sub>0-∞</sub>, CL/F, MRT, V<sub>z</sub>/F and V<sub>ss</sub>/F will not be calculated.

| Parameters | Unit | Calculation |
|---|---|---|
| C <sub>max</sub> | ng/mL | will be determined by visual inspection |
| AUC₀-∞ | ng·h/mL | $AUC_{0-\infty} = AUC_{0-t} + C_{last} / Kel$ |
| | | Clast: last measurable concentration |
| AUC%ex | % | $AUC\%_{ex} = (AUC_{0-\infty} - AUC_{0+}) / AUC_{0-\infty} \times 100$ |
| AUC <sub>0-t</sub> | ng·h/mL | will be calculated using the linear trapezoidal method and actual |
| | | times |
| | | $AUC_{0-t} = \sum_{i=1}^{n} \frac{t_i - t_{i-1}}{2} (C_{i-1} + C_i)$ |
| AUC <sub>0-24</sub> | ng∙h/mL | will be calculated using time until 24 h drug concentration |
| t <sub>max</sub> | h | Measured time of C <sub>max</sub> |
| t <sub>1/2</sub> | h | $t_{1/2}$ will be determined as: $t_{1/2} = \log_e(2)$ / Kel |
| Kel | 1/h | The exponential rate constant of the terminal phase, kel, will be |
| | | estimated by log-linear regression, if determinable. The number |
| | | of data points included in the regression will be determined by |
| | | visual inspection. Wherever possible, a minimum of 3 data points |
| | | will be used in the estimation of Kel. |
| | | During the analysis, this calculation method repeats regressions |
| | | using the last three points with non-zero concentrations, then the |
| | | last four points, last five, etc. The time of maximum concentration |
| | | (t <sub>max</sub> ) will be excluded from the estimation of K <sub>el</sub> . |
| | | Points with a value of zero for the dependent variable are |
| | | excluded. For each regression, an adjusted R <sup>2</sup> is computed |
| | | Adjusted $R^2 = 1 - \frac{(1 - R^2) \times (n - 1)}{(n - 2)}$ |
| • | | where n is the number of data points in the regression and R <sup>2</sup> is |
| | | the square of the correlation coefficient. |

| _ | | |
|---|---|---|
| | | <ul> <li>The regression with the largest adjusted R² is selected to estimate Kel, with these caveats:</li> <li>If the adjusted R² does not improve, but is within 0.0001 of the largest adjusted R² value, the regression with the larger number of points is used.</li> <li>Kel must be positive, and calculated from at least three data points.</li> </ul> |
| CL/F | L/h | $CL/F = \frac{Dose}{AUC_{0-\infty}}$ |
| MRT | h | $\begin{aligned} \text{AUMC}_{0-\infty} &= \sum_{i=1}^{n} \frac{(t_i - t_{i-1})(t_i \times C_i + t_{i-1} \times C_{i-1})}{2} + \frac{t \times C_t}{Kel} + \frac{C_t}{(Kel)^2} \\ \text{MRT}_{0-\infty} &= \frac{AUMC_{0-\infty}}{AUC_{0-\infty}} \end{aligned}$ |
| V <sub>z</sub> /F | L | $V_z/F = CL/F \times \frac{1}{Kel}$ |
| V <sub>ss</sub> /F | L | $V_{ss}/F = MRT \times CL/F$ |
| Number of Kel points | - | will be determined using number of points used in computing Kel. If Kel cannot be estimated, zero. |
| Lower Limit of Kel | h | will be determined using lower limit on time to be included in the calculation of Kel |
| Upper Limit of Kel | h | will be determined using upper limit on time to be included in the calculation of Kel |
| Ae | mg | urine concentration × urine volume |
| Ae% | % | Ae / Dose |
| CLr | L/h | $CLr = \frac{Ae}{AUC_{0-\infty}}$ |